CLINICAL TRIAL: NCT03537755
Title: The Effect of Food Marketing and Attentional Biases on Eating Behaviors in African American Adolescent Girls
Brief Title: Black Adolescent & Entertainment Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1F31MD010675-01 (NIH)
Record Dates: First submitted 2018-04-30; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Examine thoughts and behaviors

SUMMARY:
The study is being conducted to obtain adolescent girls' thoughts and opinions on relationship and communication styles are shown on television.

ELIGIBILITY:
Inclusion Criteria:

1. Female,
2. Self-identify as African American or Black,
3. 12 to 17 years of age at the start of the study,
4. Presence of obesity by virtue of a body mass index (BMI) ≥ 95th percentile for age and sex or non-overweight by virtue of a BMI of at least the5th percentile, but below the 85th percentile, for age and sex,118 and
5. English speaking.

Exclusion Criteria:

1. Reports of the presence of a major chronic medical illness: renal, hepatic, gastrointestinal, endocrinologic (e.g., Cushing syndrome, hyper- or hypothyroidism), hematological problems or pulmonary disorders (other than asthma not requiring continuous medication),
2. Individuals who self-report major depressive disorder, psychoses, current substance or alcohol use disorder, or any other psychiatric disorder that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study.
3. Current, regular use of prescription medications that affect appetite, mood, or body weight: currently prescribed serotonin re-uptake inhibitors (SSRIs), neuroleptics, tricyclics, stimulants, or any other medication known to affect appetite, mood, or body weight. Oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before the study visit,
4. Failure to provide a rating of 6 or more on at least 50% of food items on the Food Preferences Questionnaire (Appendix F); exceptions may be given for restrictions due to religious practices or food allergies, if food items can be replaced with items of equivalent macronutrient content.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Self-reported female
Study Population: Black/African American girls 12-17 years old
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Total energy consumption | Day 1
  Total energy consumption from a laboratory test meal
Macronutrient intake | Day 1
  Total energy intake from fat, sugar, and sodium

CONTACTS AND LOCATIONS:
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No